CLINICAL TRIAL: NCT03921008
Title: Induction Paclitaxel Followed by Concurrent Paclitaxel and Radiation Therapy for Cutaneous Angiosarcoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201904069
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Angiosarcoma
MeSH Terms: interventions — Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Paclitaxel and Radiation (Experimental): * All patients will receive standard of care induction chemotherapy with 6 weekly cycles of paclitaxel at 80 mg/m^2. They will then receive 6 weekly cycles of paclitaxel at 80 mg/m^2 concurrently with radiation therapy. Patients will be receiving paclitaxel as part of their routine care, but in order to participate in this study, their induction chemotherapy regimen must be paclitaxel. Radiation therapy is 50.4 Gy in 28 fractions delivered within 7 weeks. A radiation therapy boost of 10-16.2 Gy over 5-9 fractions is allowed at the discretion of the treating physician.
  * Standard of care surgery ideally within 6 weeks after completing concurrent chemotherapy and radiation therapy
  Interventions: Drug: Paclitaxel; Radiation: Radiation therapy; Procedure: Research blood draw

INTERVENTIONS:
Drug: Paclitaxel — -Commercial supply
  Other Names: Taxol
Radiation: Radiation therapy — -Patients may be treated with electrons, 3D conformal photon radiotherapy, intensity modulated photon radiotherapy (IMRT), proton radiation therapy, or a combination of these.
Procedure: Research blood draw — -Within 1 week (prior to cycle 1 of paclitaxel preferred but not required), pre-radiation therapy (any time weeks 5-7 as long as radiation therapy has not started), post-radiation therapy (day of last fraction), 14 days post-radiation therapy, and within 2 weeks post-surgery

SUMMARY:
Angiosarcoma is a rare and aggressive form of soft tissue sarcoma. Prior work demonstrates very poor outcomes, with most patients developing metastatic disease and less than 50% surviving greater than 5 years. In other soft tissue sarcomas, the use of radiotherapy and/or chemotherapy have improved progression-free survival in patients undergoing limited, organ-sparing surgeries. Taxane chemotherapy has shown efficacy in patients with metastatic angiosarcoma, but this has not been tested in patients with localized disease. This study examines the efficacy of induction paclitaxel followed by concurrent chemoradiation therapy with paclitaxel prior to curative surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cutaneous angiosarcoma.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 5 mm with CT scan or ≥ 5 mm by clinical exam at the time of diagnosis
* Currently receiving or planning to receive weekly paclitaxel for 12 weeks at 80 mg/m^2 weekly. The patient must be able to begin radiotherapy within the first 7 weeks of paclitaxel treatment.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and one month after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Patients deemed ineligible for curative therapy by the treating medical oncologist, radiation oncologist, or surgeon.
* A history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any investigational agents.
* Current central nervous system disease or distant metastatic disease not including local-regional lymph nodes or satellite lesions. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Grade 2 or greater neuropathy
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* HIV-positive patients whose CD4+ T-cell count is < 350 cells/mcL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2028-01-16 (Estimated); Study Completion 2028-01-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | At year 2 follow-up (estimated to be 2 years and 12 weeks)
  * PFS is defined as the duration of time from pathologic diagnosis to time of progression or death, whichever occurs first.
  * Progression is defined as the appearance of new angiosarcoma lesions as determined by clinical exam, radiography, and/or pathologic confirmation.

SECONDARY OUTCOMES:
Overall survival (OS) rate | At year 2 follow-up (estimated to be 2 years and 12 weeks)
  -Patients that have died from any cause will be censored from the OS rate calculation
Pathologic complete response rate (pCR) | At the time of surgery (approximately 19 weeks)
  -Defined as the lack of viable cells observed in resected tumor tissue following neoadjuvant therapy and will be determined by an experienced sarcoma pathologist
Rate of acute treatment-related grade 3 or higher toxicity defined by CTCAE version 5.0 | From start of radiation through 90 days after start of radiation
Rate of late treatment-related grade 3 or higher toxicity defined by CTCAE version 5.0 | From 91 days through year 2 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Apicelli, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy A, Gabani P, Davis EJ, Oppelt P, Merfeld E, Keedy VL, Zoberi I, Chrisinger JSA, Michalski JM, Van Tine B, Spraker MB. Concurrent paclitaxel and radiation therapy for the treatment of cutaneous angiosarcoma. Clin Transl Radiat Oncol. 2021 Jan 28;27:114-120. doi: 10.1016/j.ctro.2021.01.009. eCollection 2021 Mar. PMID 33604458
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu